CLINICAL TRIAL: NCT02951832
Title: Study About Lymphocytes Change During Menstrual Cycle in Women of Child-bearing Age
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Principal Investigator, Shihua Bao, Principal Investigator, Shanghai First Maternity and Infant Hospital
Other Study IDs: ShanghaiFMIH-RI
Record Dates: First submitted 2016-10-26; First posted 2016-11-01 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2016-11

CONDITIONS: Lymphocyte Subsets in Women of Child-bearing Age

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- observational group: Observational Study about Lymphocytes Change during Menstrual Cycle in Women of Child-bearing Age

SUMMARY:
The investigators are going to select the normal child-bearing period women as the study subjects and draw their peripheral blood to observe and analyze the change of quantity and percentage of lymphocyte subsets along with the change of menstrual cycle.

Recording their BMI\menstrual history\and childbearing history, the investigators would select 300 healthy women in 6 different age groups which are aged 20-24, aged 25-29, aged 30-34, aged35-39, aged 40-44 and aged 45-49, then draw 1-2 ml blood form their peripheral vein (adding EDTA for anti-coagulation). The investigators are going to perform routine examination on the blood samples and detect T\B\NK lymphocyte through flow cytometry (FCM), thus calculating the absolute number of every species of lymphocyte. The investigators make assessment for the cellular immune function of the women during child-bearing period via comparing distinction in percentage and absolute number of every lymphocyte subset among reproductive-age women in different ages.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20-49;
* Having a regular menstrual cycle of which the menstrual period is between day 3-7, and the period between day 25-35;
* Excluding internal and surgical disease (after having variety of physical examination such as electrocardiogram/hepatic and renal function/blood routine and urine routine).

Exclusion Criteria:

* Having experienced severe allergies, trauma history and/or operation history within 3 months;
* With a history of mental illness and/or family history of mental illness;
* Limb disabled;
* Taking medicine within one month;
* Suffering major events or having mood swings.

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy women of child-bearing age
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-03-01 (Actual); Study Completion 2017-12-10 (Estimated)

PRIMARY OUTCOMES:
the percentage of lymphocyte subsets | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tao Duan, Study Chair — Shanghai First Maternity and Infant Hospital
Locations (1):
- Shanghai first Maternity and Infant health hospital, Tong Ji University, Shanghai, China